CLINICAL TRIAL: NCT06283264
Title: Assessment of Coeliac Disease in Patients With Type 2 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Mohey Roshdy Khella, Principal investigator, Assiut University
Other Study IDs: Coeliac Disease in type2 DM
Record Dates: First submitted 2023-12-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to screen and diagnose coeliac disease in patients with type 2 diabetes and monitor the effect of gluten-free diet on the metabolic status

DETAILED DESCRIPTION:
Coeliac Disease (CD) is a chronic disease with long-term consequences if untreated . CD has been traditionally associated with autoimmune disorders as type 1 Diabetes . However, recent data suggest association with insulin resistance, metabolic syndrome and type 2 diabetes . In a recent study comparing prevalence of autoimmune markers in type 1 diabetes versus type 2, coeliac disease serologic markers were 5% versus 8.7% respectively . In a study published at Nature communication, a genetic link between Ig A levels, type 2 diabetes, and coeliac disease was found . Gluten, among other factors, is thought to play a proinflammatory role exaggerating the damage to β-cells in both type 1 and type 2 diabetes . Presentation of coeliac disease is very variable, ranging from asymptomatic, gastrointestinal symptoms, atypical symptoms, to malabsorption syndrome. Our interest of the very wide atypical presentations is poorly controlled type 2 diabetes . Moreover, it has been recently suggested that gluten-free diet improves glucose metabolism . Screening and diagnosing coeliac disease remain a highly controversial topic, especially in individuals with atypical or no symptoms. A lifelong gluten avoidance can be only justified by a solid diagnosis, achieved by histopathological diagnosis. Intestinal biopsy is invasive test with not that-accurate results. The new guidelines confirmed the accuracy of the no-biopsy approach, only in case of high-titre positive two antibody tests, as published by the European Society Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHN) . However, guidelines intended for adults still insist on biopsy for confirming final diagnosis . The only exception is the interim guidance during Corona Virus -19 ( COVID-19 ) allowing non-biopsy diagnosis with two separate serology tests . However, recent retrospective study confirmed that high titre tTG had more than 95% diagnostic rate, and duodenal biopsy was not needed . For screening, many approaches have been studied, with measuring total immunoglobulin A (IgA) and IgA tissue transglutaminase (tTG) is the obvious first choice. However, for resource-deficient economies, rapid easy cheap point-of-care tests for deamidated gliadin antibodies (DGP) have been suggested .

ELIGIBILITY:
Inclusion Criteria:

1. adult patients ≥18 years old
2. diagnosed with type 2 diabetes mellitus

Exclusion Criteria:

1. Patients already diagnosed with co-morbid autoimmune disorder
2. patient diagnosed as systemic lupus
3. diagnosed as rheumatoid arthritis
4. already diagnosed with coeliac disease

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Diabetic type 2 willing participants, after obtaining informed consent, will be subjected to full history taking, thorough clinical examination and total immunoglobulin A (IgA) and IgA tissue transglutaminase antibody (tTG-Ab). -Those with IgA deficiency or positive tTG-Ab are offered upper endoscopy for confirmation by duodenal biopsy. -Those with confirmed Coeliac Disease will be given detailed dietary advice and promoted to strictly adhere to gluten-free diet
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
1-Prevalence of coeliac disease among diabetic type 2 patient 2-its effect on glycemic control | One year
  All willing participants, after obtaining informed consent, will be subjected to full history taking thorough clinical examination and the following measures investigations:- Anthropometric measures:- weight and height will be combined to report BMI in kg/m^2). Metabolic assessment:-
  1. HbA1c
  2. Random blood glucose in mg/dl Measuring of :-
  1-total immunoglobulin A (IgA) and IgA 2- tissue transglutaminase antibody (tTG-Ab).

REFERENCES:
- [Background] Lindfors K, Ciacci C, Kurppa K, Lundin KEA, Makharia GK, Mearin ML, Murray JA, Verdu EF, Kaukinen K. Coeliac disease. Nat Rev Dis Primers. 2019 Jan 10;5(1):3. doi: 10.1038/s41572-018-0054-z. PMID 30631077
- [Background] Damms-Machado A, Louis S, Schnitzer A, Volynets V, Rings A, Basrai M, Bischoff SC. Gut permeability is related to body weight, fatty liver disease, and insulin resistance in obese individuals undergoing weight reduction. Am J Clin Nutr. 2017 Jan;105(1):127-135. doi: 10.3945/ajcn.116.131110. Epub 2016 Nov 9. PMID 28049662
- [Background] Haupt-Jorgensen M, Holm LJ, Josefsen K, Buschard K. Possible Prevention of Diabetes with a Gluten-Free Diet. Nutrients. 2018 Nov 13;10(11):1746. doi: 10.3390/nu10111746. PMID 30428550
- [Background] Liu L, Khan A, Sanchez-Rodriguez E, Zanoni F, Li Y, Steers N, Balderes O, Zhang J, Krithivasan P, LeDesma RA, Fischman C, Hebbring SJ, Harley JB, Moncrieffe H, Kottyan LC, Namjou-Khales B, Walunas TL, Knevel R, Raychaudhuri S, Karlson EW, Denny JC, Stanaway IB, Crosslin D, Rauen T, Floege J, Eitner F, Moldoveanu Z, Reily C, Knoppova B, Hall S, Sheff JT, Julian BA, Wyatt RJ, Suzuki H, Xie J, Chen N, Zhou X, Zhang H, Hammarstrom L, Viktorin A, Magnusson PKE, Shang N, Hripcsak G, Weng C, Rundek T, Elkind MSV, Oelsner EC, Barr RG, Ionita-Laza I, Novak J, Gharavi AG, Kiryluk K. Author Correction: Genetic regulation of serum IgA levels and susceptibility to common immune, infectious, kidney, and cardio-metabolic traits. Nat Commun. 2023 Feb 6;14(1):655. doi: 10.1038/s41467-023-36340-3. No abstract available. PMID 36746961
- [Background] Kizilgul M, Ozcelik O, Beysel S, Akinci H, Kan S, Ucan B, Apaydin M, Cakal E. Screening for celiac disease in poorly controlled type 2 diabetes mellitus: worth it or not? BMC Endocr Disord. 2017 Oct 6;17(1):62. doi: 10.1186/s12902-017-0212-4. PMID 28985731
- [Background] Husby S, Koletzko S, Korponay-Szabo IR, Mearin ML, Phillips A, Shamir R, Troncone R, Giersiepen K, Branski D, Catassi C, Lelgeman M, Maki M, Ribes-Koninckx C, Ventura A, Zimmer KP; ESPGHAN Working Group on Coeliac Disease Diagnosis; ESPGHAN Gastroenterology Committee; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition guidelines for the diagnosis of coeliac disease. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):136-60. doi: 10.1097/MPG.0b013e31821a23d0. PMID 22197856
- [Background] Rubio-Tapia A, Hill ID, Semrad C, Kelly CP, Greer KB, Limketkai BN, Lebwohl B. American College of Gastroenterology Guidelines Update: Diagnosis and Management of Celiac Disease. Am J Gastroenterol. 2023 Jan 1;118(1):59-76. doi: 10.14309/ajg.0000000000002075. Epub 2022 Sep 21. PMID 36602836
- [Background] Johnston RD, Chan YJ, Mubashar T, Bailey JR, Paul SP. No-biopsy pathway following the interim BSG guidance reliably diagnoses adult coeliac disease. Frontline Gastroenterol. 2020 Oct 6;13(1):73-76. doi: 10.1136/flgastro-2020-101624. eCollection 2022. PMID 34966534
- [Background] Masic M, Musil V, Petricevic Vidovic T, Sicaja E, Hojsak I, Jadresin O, Kolacek S, Misak Z. Point-of-Care Screening for Coeliac Disease in Schoolchildren Reveals Higher Disease Prevalence in Croatia. Healthcare (Basel). 2022 Dec 26;11(1):64. doi: 10.3390/healthcare11010064. PMID 36611524
- [Background] Alyafei F, Soliman A, Alkhalaf F, Sabt A, De Sanctis V, Elsayed N, Waseef R. Prevalence of beta-cell antibodies and associated autoimmune diseases in children and adolescents with type 1 diabetes (T1DM) versus type 2 diabetes (T2DM) in Qatar. Acta Biomed. 2018 May 23;89(S5):32-39. doi: 10.23750/abm.v89iS4.7359. PMID 30049930